CLINICAL TRIAL: NCT02171299
Title: Intraoperative Wound Infiltration With Local Anaesthetic in Surgical Patients; Is There Any Late Effect on the Postoperative Pain and the Requirements of Analgesia ? A Randomized Control Trial.
Brief Title: Intraoperative Local Anaesthetic and Postoperative Pain
Acronym: Pain-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Sophocles Lanitis, Dr. Sophocles Lanitis, M.D, PhD, Hellenic Red Cross Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10103
Record Dates: First submitted 2014-06-11; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Local; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervetional group (local anaesthetic) (Experimental): intraoperative wound infiltration with ropivacaine 10%.
  Interventions: Procedure: Wound infiltration with local anaesthetic; Drug: Ropivacaine
- control (no local anesthetic) (No Intervention): no infiltration of the wound with local anaesthetic

INTERVENTIONS:
Procedure: Wound infiltration with local anaesthetic
  Arms: intervetional group (local anaesthetic)
Drug: Ropivacaine
  Arms: intervetional group (local anaesthetic)

SUMMARY:
Background: Intraoperative wound infiltration with local anaesthetic is commonly used. Apart from the obvious immediate action it has been supported that a possible down regulation of pain receptors may lead to longer effects. Our aim was to compare the use of local anaesthetic versus placebo in order to assess if indeed there is a late beneficial effect.

Materials and methods: We will conduct a RCT involving 400 consecutive general surgery patients randomized in 2 groups: Group A= placebo, Group B= wound infiltration with ropivacaine 10%. We will record the preoperative and postoperative pain for the 1st week as well as the type and quantity of the analgesia used during the study period.

Hypothesis : patients who receive intraoperatively wound infiltration with local anaesthetic have lower pain during the 1st postoperative week and require less pain killers .

ELIGIBILITY:
Inclusion Criteria:

* Patients with conditions that require surgery ( general surgery)
* Must be able to comprehent the questions , fill documents, communicate well with the doctors
* Patients who will have at least one surgical incision under general or regional anaesthesia

Exclusion Criteria:

* Patients who could not comprehend well
* patients who remained intubated even for one postoperative day
* Patients who were discharged the day of the operation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Intensity of postoperative pain | six days
  the intensity of the pain will be assessed using the : The visual analogue scale (VAS) which is a psychometric response scale and the patient has to indicate a position along a continuous line between two end-points (no pain and maximum pain) and (2) the numeric rating scale (NRS) which is a segmented numeric version of the visual analog scale (VAS) in which the patient indicates the number (0-10) that best reflects the intensity of their pain. Both tests are easy to obtain, reliable, valid and can detect changes of over time

SECONDARY OUTCOMES:
Quantity and quality of the required postoperative analgesia | six days
  Nonsteroidal antiinflamatory drugs and opioids . each day the analgesia required by the patient is recorded and classified accordingly

OTHER OUTCOMES:
type of analgesia required postoperatively | six days
  whether more NSAIS or more opioids were required at any given day

CONTACTS AND LOCATIONS:
Locations (1):
- "Korgialenio-Benakio", Hellenic Red Cross Athens General Hospital, Greece, Athens, Greece

REFERENCES:
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Derived] Lanitis S, Karkoulias K, Sgourakis G, Brotzakis P, Armoutides V, Karaliotas C. The late effect of intraoperative wound infiltration with local anaesthetic in surgical patients; is there any? A randomized control trial. Int J Surg. 2015 Aug;20:35-40. doi: 10.1016/j.ijsu.2015.05.053. Epub 2015 Jun 11. PMID 26074287